CLINICAL TRIAL: NCT03682510
Title: A Randomized Clinical Trial Comparing the Efficacy of B-Lynch Transverse Compression Suture Versus a Sandwich Technique (N&H Technique) at the Time of Cesarean Delivery for Complete Placenta Previa
Brief Title: B-Lynch Transverse Compression Suture Versus a Sandwich Technique (N&H Technique) for Complete Placenta Previa
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Aswan University Hospital (Other)
Responsible Party: Principal Investigator, hany farouk, lecturer, Aswan University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: aswu/170/10/17
Record Dates: First submitted 2018-09-21; First posted 2018-09-24 (Actual); Last update posted 2018-12-13 (Actual); Status verified 2018-12

CONDITIONS: Cesarean Section Complications
Keywords: placenta previa; transverse b lynch suture; N&H sandwich technique
MeSH Terms: conditions — Placenta Previa

STUDY DESIGN:
Intervention Model Description: The participants who fulfilled the eligibility criteria were explained about the study with the beneficial and possible adverse effects of lidocaine. Informed consent was obtained from them after that participant were randomized into 3 groups: group 1 [N&H technique], group 2 [N&H technique] and group 3 stepwise devascularization
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- stepwise devascularization (Active Comparator): routine stepwise devascularization
  Interventions: Procedure: stepwise devascularization
- B-Lynch Transverse Compression Suture (Active Comparator): After acceptable control of bleeding from the placental bed, uses the suture material 1 VICRYL with a 70mm ½ circle needle mounted on a 90 cms VICRYL suture. We use the needle blunt ended to puncture the uterus 3 cms above the upper margin of the incision posteriorly and behind the vascular bundle.
  The needle is retrieved through the cavity of the uterus and pulled inferiorly with the suture material lying on the posterior wall of the uterine cavity. The needle then perforates the posterior wall of the uterus 3 cms below the inferior margin of the Caesarean incision and exists behind the vascular bundle of the same side of the uterus retrieved and runs on the surface of the lower segment below the incision margin parallel to it and taking a 1 cm bite of tissue for stabilization running to the other side.
  Interventions: Procedure: B-Lynch Transverse Compression Suture group
- N&H technique (Experimental): In the N&H group, double uterine compression suture at the lower uterine segment with inflated Foley's catheter balloon tamponade. As follow:
  (i) 100-cm Vicryl no. 1 was thrown to form two nearly equal parts (each 50 cm) on a blunt semicircular 70-mm needle, the curve of the needle was straightened.
  (ii) The needle transfixed the right side of the uterine wall from anterior to posterior, about 2 cm below the hysterotomy incises posterior, then the needle transfixed the left side of the uterine wall from posterior to anterior, about 2 cm below the hysterotomy incision.
  Interventions: Procedure: N&H sandwich technique

INTERVENTIONS:
Procedure: stepwise devascularization — stepwise devascularization begins with suture the placenta bed through uterine artery ligation, internal iliac artery ligation etc
  Arms: stepwise devascularization
Procedure: B-Lynch Transverse Compression Suture group — After acceptable control of bleeding from the placental bed, uses the suture material 1 VICRYL with a 70mm ½ circle needle mounted on a 90 cms VICRYL suture. We use the needle blunt ended to puncture the uterus 3 cms above the upper margin of the incision posteriorly and behind the vascular bundle.
  The needle is retrieved through the cavity of the uterus and pulled inferiorly with the suture material lying on the posterior wall of the uterine cavity. The needle then perforates the posterior wall of the uterus 3 cms below the inferior margin of the Caesarean incision and exists behind the vascular bundle of the same side of the uterus retrieved and runs on the surface of the lower segment below the incision margin parallel to it and taking a 1 cm bite of tissue for stabilization running to the other side. After encircling the para-uterine vasculature, the needle then perforates the posterior side of the uterus behind the vascular bundle entering the uterine cavity.
  Arms: B-Lynch Transverse Compression Suture
Procedure: N&H sandwich technique — In the N&H group, double uterine compression suture at the lower uterine segment with inflated Foley's catheter balloon tamponade.
  Arms: N&H technique

SUMMARY:
Obstetric hemorrhage is estimated to be responsible for about 30% of all maternal deaths and is the leading direct etiology of maternal mortality worldwide . Especially in developing countries, hemorrhage is by far the leading cause of mortality and morbidity, with 140,000 women dying of PPH worldwide each year, which equates to 1 death every 4 min . The United Nations Millennium Development Fifth Goal, to reduce 75 % of maternal mortality by 2015 that not reached yet, cannot be held without significant improvements in postpartum hemorrhage (PPH) related mortality.

Placenta previa (PP) is an obstetric condition that is closely linked with potentially life-threatening hemorrhage with varied incidence approximately four or five per 1000 pregnancies. Placenta previa is diagnosed when the placenta obstructs part or all the cervical os during antenatal ultrasonography. Placenta previa may be subclassified using ultrasound scan to be "major or complete" (implanted across the cervix) or "minor" (not implanted across the cervix).

Currently, there is a dramatic increase in the incidence of placenta previa due to the increasing rate of cesarean delivery combined with increasing maternal age (6) It is considered one of the causes of the increased need for blood transfusion and cesarean hysterectomy.

Various conservative measures have been developed to avoid hysterectomy and preserve fertility in patients with PP. Bilateral Uterine artery ligation (BUAL) is one of the reported surgical procedures carried out in these cases as it is easy and quick. It can be used alone or with adjunctive measures with a fair success rate. The aim is to reduce the blood supply to the uterus and to prevent PPH.

There are a few methods to prevent and treat placenta previa bleeding immediately after cesarean delivery and control intra-operative bleeding during the cesarean operation. A safe intra-operative maneuver to arrest bleeding due to placenta previa is required. However, there is no gold standard treatment of placenta previa hemorrhage. The aims of the study to assess the effect of the novel sandwich technique for the control of hemorrhage during cesarean section due to placenta previa (double Transverse Compression Suture at the lower uterine segment plus Intrauterine inflated Foley's Catheter Balloon, (N&H technique) on control of massive bleeding due to central placenta previa in comparison with B-Lynch Transverse Compression Suture.

DETAILED DESCRIPTION:
All participants will undergo a detailed history, general, abdominal and vaginal examinations, body mass index (BMI) was calculated and pelvic ultrasound examination was undertaken for all participants. The participants who fulfilled the eligibility criteria were explained about the study with the beneficial and possible adverse effects of lidocaine. Informed consent was obtained from them after that participant will be randomized into 3 groups: group 1 [N&H technique], group 2 [N&H technique] and group (3) stepwise devascularization Eligible participants will be allocated to one of 3 groups after induction of general anesthesia and prior to the operation and before skin incision. The abdomen was exposed through Pfannenstiel incision, after skin incision, the subcutaneous fat and abdominal fascia were opened crosswise, and the rectus muscle was opened on the midline, the parietal peritoneum was opened longitudinally, the visceral peritoneum was opened transversely and dissected downwards with the bladder and kept against symphysis pubis by a Doyen retractor, followed by transverse incision of the uterus at the upper border of the placenta to avoid transplacental incision which provokes severe bleeding . The fetus was delivered.

20 IU oxytocin was given IV infusion after IIAL to prevent premature separation of placenta which provoked severe bleeding then placenta delivery was done.

In the B-Lynch Transverse Compression Suture group, After acceptable control of bleeding from the placental bed, uses the suture material 1 VICRYL with a 70mm ½ circle needle mounted on a 90 cms VICRYL suture. We use the needle blunt ended to puncture the uterus 3 cms above the upper margin of the incision posteriorly and behind the vascular bundle.

The needle is retrieved through the cavity of the uterus and pulled inferiorly with the suture material lying on the posterior wall of the uterine cavity. The needle then perforates the posterior wall of the uterus 3 cms below the inferior margin of the Caesarean incision and exists behind the vascular bundle of the same side of the uterus retrieved and runs on the surface of the lower segment below the incision margin parallel to it and taking a 1 cm bite of tissue for stabilization running to the other side. After encircling the para-uterine vasculature, the needle then perforates the posterior side of the uterus behind the vascular bundle entering the uterine cavity. The suture can lie freely on the posterior wall of the uterine cavity and exists 3 cms above the upper margin of the Caesarean incision. It exits posteriorly and behind the vascular bundle to meet the suture from the other side.

It is essential that the ureters are identified by palpation or visual observation after the bladder is displaced inferiorly and held by traction. Any observed bleeding should be dealt with in the usual way. At the end of the suture application and before tying the knots, the lower segment is compressed again transversely whilst the suture is held taut to ensure that bleeding has ceased by swabbing the vagina again.

A wide pore drain was then inserted in the Douglas pouch, and the abdominal wall was repaired. In the case of conservative treatment protocol failure, cesarean hysterectomy was performed

ELIGIBILITY:
Inclusion Criteria:

* all pregnant women with a single term fetus scheduled for elective CS for complete PP and invited them to participate in the study. PP was defined as a placenta completely covering the cervical os in ultrasound examination

Exclusion Criteria:

* 1-Patients with the cardiac, hepatic, renal or thromboembolic disease. 2- patients with the high possibility of the morbid adherent placenta. 3-known coagulopathy and 4- those presented with severe antepartum hemorrhage will be excluded

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — pregnant women need a cesarean section for placenta previa
Enrollment: 35 (Estimated)
Dates: Start 2018-10-31 (Actual); Primary Completion 2021-09-30 (Estimated); Study Completion 2022-01-01 (Estimated)

PRIMARY OUTCOMES:
estimation of intraoperative blood loss (ml). | during the operation
  Intraoperative blood loss was measured suction bottle and the difference in weight (in grams) between the dry and the soaked operation sheets and towels (1 gram = 1 ml.). Post-operative blood loss was measured through intraperitoneal suction drain which measured every 12 hours and on removing the drain. After that, the total blood loss was calculated by the addition of intraoperative and postoperative blood loss.and vaginal bleeding

SECONDARY OUTCOMES:
need for blood transfusion | 24 hours postoperative
  need for blood transfusion
Hemoglobin concentration | ist 24 hours postoperative
  pre and postoperative hemoglobin estimation
need of extra surgical maneuvers | during operation
  internal iliac ligation or hysterectomy

CONTACTS AND LOCATIONS:
Locations (1):
- AswanUH, Aswān, Egypt

IPD SHARING:
Plan to Share IPD: Undecided